CLINICAL TRIAL: NCT02978079
Title: Automated Pupillometry for the Diagnosis of Horner's Syndrome in Acute Stroke Patients Due to Carotid Artery Dissection
Brief Title: Pupillometry in Horner's Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Konrad Peter Weber, Principal Investigator, University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KEK-Nr. 2016-02151
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Horner's Syndrome; Stroke; Dissection Carotid Artery
MeSH Terms: conditions — Horner Syndrome; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pupillometry in stroke patients (Experimental): All eligible patients will undergo pupillometry test for the finding of Horner's syndrome
  Interventions: Device: Automated pupillometry

INTERVENTIONS:
Device: Automated pupillometry — Automated pupillometry will be performed in patients with acute stroke with the intention of diagnosing Horner's syndrome

SUMMARY:
Horner's syndrome (HS) is a result of interruption of the sympathetic innervation to the eye and ocular adnexa, which can occur due to carotid artery dissection (CAD), along which the sympathetic nerve fibers travel to reach the eye. Dissection of the carotid artery is one of the etiologies for ischemic stroke in young patients.

In our current study, we will explore the diagnostic accuracy of automated binocular pupillometry in the diagnosis or HS, and its potential in identifying dissection of the carotid artery in patients of young age who suffer ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adults 60 years of age or younger
* Acute stroke (less than 72 hours from admission)
* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Ability to understand the study information and consent form

Exclusion Criteria:

* known history of HS
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Medications affecting pupillary response
* History of ocular surgery affecting the pupil

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Finding of pupillary dilation lag using pupillometry in patients with acute stroke due to carotid artery dissection | 1 day of initial visit

CONTACTS AND LOCATIONS:
Overall Officials: Konrad P Weber, MD, Principal Investigator — Ophthalmology Department, University Hospital Zurich
Locations (1):
- Ophthalmology Department, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No